CLINICAL TRIAL: NCT00778180
Title: A Study to Compare the Relative Bioavailability of Ranbaxy and Aventis Formulations of Furosemide 80 mg Tablets in Healthy Adult Volunteers Under Fasted Condition.
Brief Title: Bioequivalence Study of Furosemide 80mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10540344
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence furosemide 80 mg tablets
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): furosemide 80 mg tablets of Ranbaxy
  Interventions: Drug: furosemide 80 mg tablets
- 2 (Active Comparator): Lasix® (furosemide) 80 mg tablets
  Interventions: Drug: furosemide 80 mg tablets

INTERVENTIONS:
Drug: furosemide 80 mg tablets

SUMMARY:
The purpose of this study was to evaluate the relative bioavailability of the test formulation of furosemide 80 mg tablets (Ohm Laboratories, Inc.) with an already marketed reference formulation Lasix® (furosemide) 80 mg tablets (Aventis Pharmaceuticals NJ) under fasted conditions in healthy adult human subjects

DETAILED DESCRIPTION:
This randomized, single-dose, two-way, crossover study was conducted to compare the relative bioavailability of two formulations of 80 mg furosemide tablets under fasted conditions. The study was conducted with 44 (39 completing) healthy adults in accordance with protocol. In each study period, a single 80 mg dose was administered to the subjects following an overnight fast. The test formulation was furosemide 80 mg tablet (Ohm Laboratories, Inc.), and the reference formulation was Lasix® (furosemide) 80 mg tablet (Aventis Pharmaceuticals NJ). The subjects received the test product in one study period and the reference product in the other period; the order of administration was according to the dosing randomization schedule. There was a 7-day interval between treatments.

Blood samples were collected pre-dose and at intervals over 12 hours after each dose. The plasma samples for all subjects completing both periods of the study were sent to BA Research, 10550 Rockley Road, Suite 150, Houston, Texas 77099, Telephone: 281-495-6996, Fax 281-575-6996 for determination of furosemide plasma concentration.

Statistical analysis was performed at Ba Research, 2591 Sam Bass Road, Round Rock, TX 78681, Telephone 512-388-4554, Fax 512-388-4550.

A total of 44 subjects were randomized to receive single oral dose of 80 mg furosemide tablets and 39 subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females aged 18 years of age or older with a body mass index (BMI) in the range 18-30 kg/m2 inclusive, measured according to Novum Standard Operating Procedures.

  * Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
  * Signed and dated informed consent form, which meets all criteria of current FDA regulations.
  * Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable method of contraception (e.g. condom with spermicide, IUD, hormonal contraceptives) for at least 30 days prior to dosing and during the duration of the study. All females in the study will have pregnancy tests performed at screening at check-in each study period.

Exclusion Criteria:

* Females who are pregnant, lactating or likely to become pregnant during the study.

  * History of allergy or sensitivity to Furosemide, other thiazide, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
  * Significant history or current evidence of chronic infectious disease, system disorder or organ dysfunction. Subjects with any history of hepatic disease or pancreatitis will be excluded.
  * Presence of gastrointestinal disease or history of malabsorption within the last year.
  * History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
  * Presence of a medical condition requiring regular treatment with prescription drugs.
  * Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing.
  * Receipt of any drug as part of a research study within 30 days prior to dosing.
  * Drug or alcohol addiction requiring treatment in the past 12 months.
  * Donation or significant loss of whole blood (480 ml or more) with/n 30 days or plasma within 14 days prior to dosing.
  * Positive test results for HIV, Hepatitis B surface antigen or Hepatitis C ant/body.
  * Positive test results for drugs of abuse at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-10; Primary Completion 2005-10 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html